CLINICAL TRIAL: NCT00462527
Title: Cystatin C as a Marker for Detecting Early Renal Dysfunction in a Pediatric Emergency Department
Acronym: CARING
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Responsible Party: Ronald Tam, MD, Staff Pediatrician, Children's Hospital of Eastern Ontario
Other Study IDs: PSI 06-49
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2007-09

CONDITIONS: Acute Renal Failure; Gastroenteritis; Dehydration
Keywords: Cystatin C; Acute renal failure; Gastroenteritis; Dehydration
MeSH Terms: conditions — Acute Kidney Injury; Gastroenteritis; Dehydration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Acute renal failure (ARF) is a rare but serious complication of gastroenteritis and dehydration, the most common reason for pediatric emergency visits. Renal function is determined by the glomerular filtration rate (GFR). Serum creatinine, the current marker of GFR, is insensitive and a late marker of ARF. Unfortunately, "gold standard" methods for measurement of GFR are impractical in the emergency setting. Recently, cystatin C (CysC) was introduced as superior marker for the measurement of GFR, particularly in children. A single random blood sample allows for accurate determination of GFR in the so-called "creatinine-blind" range and independent of the body composition. There is growing evidence that the determination of serum CysC concentration can detect ARF in adults earlier than serum creatinine or urinary fractional sodium excretion. No studies have examined this marker for the early detection of ARF in children at risk. We therefore propose a prospective study that compares CysC with other biomarkers of renal dysfunction for the early detection of ARF in children with dehydration due to gastroenteritis. Patients with minor trauma and a minimal likelihood of ARF will serve as a control. This study may establish CysC as an accurate and cost-effective marker for identifying patients at risk.

DETAILED DESCRIPTION:
* Rationale and hypotheses: Acute renal failure is a relatively rare but serious illness in children. Early detection is important in preventing life threatening complications that can arise from acute renal failure. Presently, most methods of determining renal function are either too cumbersome, too invasion or too unreliable to be used in children. Current evidence has shown that serum cystatin C is more precise and cost-effective in determining renal function. Our objective is to compare serum cystatin C with other biomarkers as an early diagnostic detection for renal dysfunction in children with acute renal failure in an emergency setting.
* Study design and methods: This is a prospective double cohort control study to compare the serum creatinine and serum cystatin C in detecting early renal dysfunction in children presenting to the emergency department. The study will be conducted in CHEO emergency department. A study nurse will identify eligible patients and discuss whether to approach the families with either the bedside nurse or attending physician before meeting them. Interested families are than given an explanation of our study. Once written consent is obtained, a copy will be given to the family. Additional tests will than be requested from blood and urine samples of the patients. Only patients that already require an intravenous needling are eligible for this study. No additional needling is therefore needed as part of this study. Urine sample will only be obtained through bad or voiding samples. No catheter urine samples will be requested as part of this study.
* Subject selection: Our target population are patients presenting to the CHEO emergency department with the diagnoses of gastroenteritis and dehydration, and requiring intravenous rehydration. Our control group are patients with traumatic injury requiring conscious sedation and intravenous access. We will exclude patients who are known to have underlying kidney diseases, renal transplantation, thyroid dysfunction, chronic systematic steroid uses, genitourinary trauma and patients transferred from another hospitals for ongoing assessment and treatment.
* Specify the number of participants drawn from CHEO and other centres: CHEO is the only designated centre for the study. 464 patients will be recruited to complete the study, 232 in each arm.
* Delineate the outcomes to be measured and analyzed: The primary outcome measures are to compare the sensitivity and the timing of detecting early renal dysfunction using either serum creatinine or serum cystatin C in the paediatric emergency setting. Our secondary outcome measures are to compare serum cystatin C to other surrogate renal markers for acute renal failure. Other renal markers include calculated Schwartz glomerular filtration rate, urine microprotein excretion, fractional excretions of sodium and urea, serum sodium, chloride, bicarbonate, urine Na/K ratio and regular urinalysis. Additional analysis will be conducted on the comparison of fractional excretion of urea to fractional excretion of sodium as an earlier marker of dehydration in children.
* Anticipated benefits/harms and how these will be addressed: Only patients who already require needling as part of their hospital care are eligible for the study. No additional needling is therefore requested. Additional tests will be requested that would otherwise not be part of the routine care of these patients. It is therefore possible that a kidney disorder will be identified in a child who was not yet diagnosed with this disease. We will discuss this possibility with the family before enrollment of the patient. All major abnormalities will be followed by both the attending physician and the principle investigators of the study and appropriate care will apply. We do not intervene with the ongoing care of the patients while the patients remain in hospital. The study will terminate when patients are discharged from the hospital.
* Data fields (if any) to be abstracted from the patient's health record: We will record patient's CHEO medical record number for the purpose of retrieving laboratory data; date of birth; biometric measurement (height, weight and sex). No other identifiable information will be record on the data sheet. No individual information will be used for publication or presentation.

Informed consent documents and any advertisement notices must be appended to the application. Both English and French versions of the consent forms and information sheets are enclosed with this application.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 18 years old presented with acute gastroenteritis with dehydration, requiring intravenous fluid rehydration

Exclusion Criteria:

* Children with known renal diseases, renal transplantation, thyroid dysfunction, chronic systematic steroid uses, genitourinary trauma
* Children transferred from another facility for ongoing assessment and treatment
* Children under legal custody
* Voluntary refusal

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Children less than 18 years old who visit the treating pediatric emergency department.
  Gastro cohort: children suffer acute gastroenteritis with signs of dehydration and require intravenous fluid rehydration Injury cohort: children suffer musculoskeletal injury that require intravenous sedation for the repair
Sampling Method: Non-Probability Sample
Enrollment: 464 (Estimated)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Tam, MD, Principal Investigator — Children's Hospital of Eastern Ontario
Locations (1):
- Department of Pediatric Emergency, Children's Hospital of Eastern Ontario, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Tam RK, Wong H, Plint A, Lepage N, Filler G. Comparison of clinical and biochemical markers of dehydration with the clinical dehydration scale in children: a case comparison trial. BMC Pediatr. 2014 Jun 16;14:149. doi: 10.1186/1471-2431-14-149. PMID 24935348